CLINICAL TRIAL: NCT00227279
Title: A Randomized, Parallel-group, Double-blind, Placebo-controlled Phase III Trial Assessing the Efficacy and Safety of ALK Grass Tablet in Subjects With Seasonal Grass Pollen Induced Rhinoconjunctivitis
Brief Title: A Trial of the ALK Grass Tablet in Subjects With Hayfever
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GT-08; NCT00146991 (obsolete NCT alias)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Allergy
Keywords: Grass pollen allergy; Hayfever; Allergen immunotherapy; Specific immunotherapy
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: ALK Grass tablet
- 2 (Placebo Comparator)
  Interventions: Biological: ALK Grass tablet

INTERVENTIONS:
Biological: ALK Grass tablet — Tablets, 75,000 SQ-T or matching placebo. Daily administration for 3 years

SUMMARY:
This trial is performed to assess the efficacy and safety of the ALK Grass tablet for treatment of grass pollen induced rhinoconjunctivitis (hayfever).

ELIGIBILITY:
Eligibility Criteria:

* A history of grass pollen induced rhinoconjunctivitis
* Positive skin prick test to grass
* Positive specific IgE to grass

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2004-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Recording of rhinoconjunctivitis symptoms | Daily recordings during the entire grass pollen seasons 2007, 2008 and 2009
Recording of use of rescue medication | Daily recordings during the entire grass pollen seasons 2007, 2008 and 2009

SECONDARY OUTCOMES:
Quality of life | Weekly recordings during the entire grass pollen seasons 2007, 2008 and 2009

CONTACTS AND LOCATIONS:
Overall Officials: Bente Tholstrup, MSc, Study Director — ALK-Abello A/S
Locations (1):
- Lungemedicinsk Forskningsafdeling, Aarhus Kommunehospital, Aarhus C, Denmark

REFERENCES:
- [Result] Dahl R, Kapp A, Colombo G, de Monchy JG, Rak S, Emminger W, Rivas MF, Ribel M, Durham SR. Efficacy and safety of sublingual immunotherapy with grass allergen tablets for seasonal allergic rhinoconjunctivitis. J Allergy Clin Immunol. 2006 Aug;118(2):434-40. doi: 10.1016/j.jaci.2006.05.003. PMID 16890769
- [Result] Durham SR, Riis B. Grass allergen tablet immunotherapy relieves individual seasonal eye and nasal symptoms, including nasal blockage. Allergy. 2007 Aug;62(8):954-7. doi: 10.1111/j.1398-9995.2007.01402.x. PMID 17620075
- [Result] Calderon MA, Birk AO, Andersen JS, Durham SR. Prolonged preseasonal treatment phase with Grazax sublingual immunotherapy increases clinical efficacy. Allergy. 2007 Aug;62(8):958-61. doi: 10.1111/j.1398-9995.2007.01416.x. PMID 17620076
- [Result] Dahl R, Kapp A, Colombo G, de Monchy JG, Rak S, Emminger W, Riis B, Gronager PM, Durham SR. Sublingual grass allergen tablet immunotherapy provides sustained clinical benefit with progressive immunologic changes over 2 years. J Allergy Clin Immunol. 2008 Feb;121(2):512-518.e2. doi: 10.1016/j.jaci.2007.10.039. Epub 2007 Dec 26. PMID 18155284